CLINICAL TRIAL: NCT04430439
Title: Postprandial Response to Emotion-Diet Interactions in Pregnancy
Brief Title: Emotion-Diet Interactions in Pregnancy
Acronym: PREDIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Karen Lindsay, Assistant Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20205914; R00HD096109 (NIH)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related; Stress, Psychological; Glucose Intolerance During Pregnancy; Emotional Stress; Postprandial Hyperglycemia; Insulin Sensitivity/Resistance
MeSH Terms: conditions — Stress, Psychological; Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be first randomized in a parallel design to meal type (low vs high GI). Within the meal arms, participants will be randomized in a cross-over design to undergo the lab-based stress and non-stress tasks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial stress (Experimental): Participants will complete the Trier Social Stress Test (TSST) immediately following consumption of their assigned meal type (low or high GI).
  Interventions: Behavioral: Psychosocial stress
- Control non-stress (Active Comparator): Participants will complete a non-stress relaxed task immediately following consumption of their assigned meal type (low or high GI).
  Interventions: Behavioral: Control non-stress

INTERVENTIONS:
Behavioral: Psychosocial stress — The TSST is a 15 minute standardized lab-based challenge task that involves speech preparation, speech delivery while being evaluated by strangers and video taped, and complex mental arithmetic with critiques if errors are made.
  Arms: Psychosocial stress
Behavioral: Control non-stress — Participants will have a relaxed 15 minute conversation with a familiar research team member.
  Arms: Control non-stress

SUMMARY:
This study will investigate how maternal emotional state following a controlled stress exposure in pregnancy influences blood glucose and insulin levels after eating a standardized meal, and whether the effects of emotional state on blood glucose and insulin is different after eating a healthy meal (low GI) compared to a less healthy meal (high GI).

DETAILED DESCRIPTION:
Maternal glucose-insulin homeostasis in pregnancy represents one of the most important physiological processes for maternal and child health outcomes. Although maternal diet is a key regulator of this process, its effects vary widely across individuals. Maternal stress could represent a moderator of considerable importance in this regard, yet little is known about the effects of stress on glycemic control in pregnancy and whether the effects of stress may vary as a function of diet quality. This project will investigate the effects of acute psychosocial stress exposure on the postprandial metabolic response to a meal of varying glycemic index (GI) among women with overweight/obesity in mid-pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* English and/or Spanish speaking
* 18-22 week's gestation
* Pre-pregnancy BMI 25.0-39.9 kg/m2
* Singleton, intrauterine pregnancy
* Non-smoker
* Non-diabetic and normal result on a random peripheral blood glucose test at the screening visit (<200 mg/dl)

Exclusion Criteria:

* Non-fluency in English or Spanish
* BMI <25.0 or ≥40.0 kg/m2
* >22 week's gestation
* multiple pregnancy
* current smoker
* present/prior obstetric conditions (preeclampsia, infections, placental abnormalities, uterine anomalies, congenital malformations, fetal chromosomal abnormalities)
* presence of any conditions that may dysregulate neuroendocrine, metabolic or cardiovascular function, such as diabetes, hepatic, renal, or autoimmune disorders
* current psychiatric disorders or undergoing treatment/taking psychiatric medications
* use of systemic/frequent corticosteroids or thyroid, lipid-lowering or anti-diabetic medications
* gestational diabetes mellitus or raised glucose result detected on the screening visit
* unwilling to eat the standard breakfast meal at each laboratory visit

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - UCI Medical Center, University of California, Irvine, Orange, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between May 2021 and February 2024, primarily from prenatal clinics affiliated with the UCI medical center. Some participants from non-UCI clinics were recruited by circulating study flyers by university-wide email and sharing with local business/non-profit organizations.
Pre-assignment Details: Upon confirmation of eligibility and completing the consent visit, participants were immediately assigned to the low or high GI meal groups and randomized to the order of their stress or non-stress lab visits.
Groups:
- Low GI Meal - Stress, Then No Stress: Participants assigned to this group consumed a low glycemic index breakfast at both study visits (nutrition shake high in fiber with minimal added sugars). On the first study visit they were exposed to the standardized stress task (TSST), followed by a 1-2 weeks washout period, followed by their second study visit with the standardized non-stress task. At both study visits, blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- Low GI Meal - No Stress, Then Stress: Participants assigned to this group consumed a low glycemic index breakfast at both study visits (nutrition shake high in fiber with minimal added sugars). On the first study visit they were exposed to the standardized non-stress task, followed by a 1-2 week washout period, followed by their second study visit with the standardized stress task (TSST). At both study visits, blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- High GI Meal - Stress, Then No Stress: Participants assigned to this group consumed a high glycemic index breakfast at both study visits (nutrition shake high in added sugars and low in fiber, plus a portion of apple sauce). On the first study visit they were exposed to the standardized stress task (TSST), followed by a 1-2 week washout period, followed by their second study visit with the standardized non-stress task. At both study visits, blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- High GI Meal - No Stress, Then Stress: Participants assigned to this group consumed a high glycemic index breakfast at both study visits (nutrition shake high in added sugars and low in fiber, plus a portion of apple sauce). On the first study visit they were exposed to the standardized non-stress task, followed by a 1-2 week washout period, followed by their second study visit with the standardized stress task (TSST). At both study visits, blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
Period: First Intervention
Arm/Group | Low GI Meal - Stress, Then No Stress | Low GI Meal - No Stress, Then Stress | High GI Meal - Stress, Then No Stress | High GI Meal - No Stress, Then Stress
Started | 30 | 27 | 22 | 34
Completed | 26 | 22 | 20 | 28
Not Completed | 4 | 5 | 2 | 6
Period: Second Intervention
Arm/Group | Low GI Meal - Stress, Then No Stress | Low GI Meal - No Stress, Then Stress | High GI Meal - Stress, Then No Stress | High GI Meal - No Stress, Then Stress
Started | 26 | 22 | 20 | 28
Completed | 22 | 15 | 20 | 23
Not Completed | 4 | 7 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Population for baseline analysis matches the number of participants who started the first intervention in Participant Flow section
Groups:
- Low GI Meal: Participants assigned to this group consumed a low glycemic index breakfast at both study visits (nutrition shake high in fiber with minimal added sugars). Blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- High GI Meal: Participants assigned to this group consumed a high glycemic index breakfast at both study visits (nutrition shake high in added sugars plus a portion of apple sauce). Blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- Total: Total of all reporting groups
Arm/Group | Low GI Meal | High GI Meal | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.60 (5.45) | 27.96 (5.41) | 28.28 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 48 | 92
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 9 | 14
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 19 | 35
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 25 | 23 | 48
Pre-pregnancy body mass index (ppBMI) [Mean (Standard Deviation); unit: Kg/m^2] — Computed based on self-reported pre-pregnancy weight and height
  Kg/m^2 | 30.34 (4.06) | 30.86 (3.83) | 30.6 (3.94)

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glycemic Response With Stress Exposure
Description: Glycemic response (area-under-the-curve of glucose) to the assigned meal type during the visit with the psychosocial stress task (TSST)
Time Frame: 2 weeks
Population: 15 participants only completed the first lab visit and missed the second visit. Of those, 11 were assigned to undergo the stress task at visit 2 and thus are missing data for the present outcome.
  Among those who did complete the visit with the stress task, some participants had insufficient blood sample collections at fasting or later timepoints, such that glucose values were missing and glucose AUC could not be computed.
Measure: Mean (Standard Deviation); unit: mg/dl * minutes
Groups:
- Low GI Meal: Participants assigned to this group consumed a low glycemic index breakfast at both study visits (i.e. before the standardized stress task during one visit and before non-stress task during the other visit). Blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
- High GI Meal: Participants assigned to this group consumed a high glycemic index breakfast at both study visits (i.e. before the standardized stress task during one visit and before non-stress task during the other visit). Blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
Arm/Group | Low GI Meal | High GI Meal
Number analyzed (Participants) | 37 | 38
mg/dl * minutes | 12998.83 (3507.22) | 12833.69 (4643.66)

2. Primary Outcome: Postprandial Glycemic Response Without Stress Exposure
Description: Glycemic response (glucose area-under-the-curve) to the assigned meal type during the visit with the non-stress control condition
Time Frame: 2 weeks
Population: 15 participants only completed lab visit 1 and missed lab visit 2. Of those, 3 were assigned to undergo the non-stress task on visit 2 and thus are missing data for this analysis.
  Some participants had insufficient blood sample collections at fasting or later timepoints, such that glucose values were missing and glucose AUC could not be computed.
Measure: Mean (Standard Deviation); unit: mg/dl * minutes
Arm/Group | Low GI Meal | High GI Meal
Number analyzed (Participants) | 38 | 45
mg/dl * minutes | 12754.18 (3028.18) | 13099.27 (4038.88)

3. Secondary Outcome: Postprandial Insulin Response With Stress Exposure
Description: Insulin response (area-under-the-curve) to the assigned meal type during the visit with the standardized stress task
Time Frame: 2 weeks
Population: 15 participants only completed the first lab visit and missed the second visit. Of those, 11 were assigned to undergo the stress task at visit 2 and thus are missing data for the present outcome.
  Among those who did complete the visit with the stress task, some participants had insufficient blood sample collections at fasting or later timepoints, such that insulin values were missing and insulin AUC could not be computed.
Measure: Mean (Standard Deviation); unit: uU/ml * minutes
Arm/Group | Low GI Meal | High GI Meal
Number analyzed (Participants) | 35 | 34
uU/ml * minutes | 7142.74 (3329.37) | 10782.48 (3704.12)

4. Secondary Outcome: Postprandial Insulin Response Without Stress Exposure
Description: Insulin response (area-under-the-curve) to the assigned meal type during the visit with the non-stress control condition
Time Frame: 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: uU/ml * minutes
Groups:
- High GI Meal: Participants assigned to this group consumed a high glycemic index breakfast at both study visits (nutrition shake high in added sugars and low in fiber, plus a portion of apple sauce). Blood and saliva samples were collected at baseline (fasting) immediately before consuming the meal, and then at 7 postprandial defined timepoints until 2.5 hours.
Arm/Group | Low GI Meal | High GI Meal
Number analyzed (Participants) | 39 | 40
uU/ml * minutes | 6791.51 (2865.53) | 11027.89 (3437.65)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 8 weeks
Groups:
- Psychosocial Stress: Participants will complete the Trier Social Stress Test (TSST) immediately following consumption of their assigned meal type (low or high GI). All participants also complete the non-stress task following consumption of their assigned meal type on a different day in a crossover design.
Arm/Group | Psychosocial Stress
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 0/113

LIMITATIONS AND CAVEATS:
Could not obtain an assay to test free fatty acids from plasma samples so we were unable to fulfill the aim of assessing the impact of stress exposure on postprandial fatty acid response to the meals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT04430439/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT04430439/SAP_001.pdf